CLINICAL TRIAL: NCT02205528
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Phase 2a Study With an Open-Label Active Group to Assess the Efficacy and Safety of Once-Daily NNC0090-2746 in Type 2 Diabetic Patients Inadequately Controlled With Metformin
Brief Title: A Study of Once-Daily NNC0090-2746 in Participants With Type 2 Diabetes Inadequately Controlled With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9709-4336; U1111-1189-5627 (Other: World Health Organization (WHO))
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Diabetes; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Treatment Period: Placebo QD (Placebo Comparator): Participants will receive daily SC placebo injections during the 12-week, double-blind treatment period.
  Interventions: Drug: Metformin; Drug: Placebo
- Treatment Period: NNC0090-2746 QD (Experimental): Participants will receive daily 1.8-mg SC injections of NNC0090-2746 during the 12-week, double-blind treatment period.
  Interventions: Drug: Metformin; Drug: NNC0090-2746
- Treatment Period: Liraglutide QD (Active Comparator): Participants will receive open-label liraglutide via SC injection during the 12-week treatment period. The dose scheme will be as follows: 0.6 milligrams (mg) each day during Week 1, followed by 1.2 mg each day during Week 2, and 1.8 mg each day from Weeks 3 to 12.
  Interventions: Drug: Liraglutide; Drug: Metformin

INTERVENTIONS:
Drug: Liraglutide — Liraglutide will be self-administered daily via SC injection according to manufacturer specifications.
  Arms: Treatment Period: Liraglutide QD
Drug: Metformin — Metformin hydrochloride immediate- or extended-release oral tablets will be supplied by the participant or investigational site as standard-of-care treatment beginning at least 8 weeks prior to randomization and throughout the 12-week treatment period. Metformin will also be continued during the 4-week follow-up. Dose selection will be based upon manufacturer specifications.
Drug: Placebo — Matching placebo to NNC0090-2746 will be self-administered daily via SC injection.
  Arms: Treatment Period: Placebo QD
Drug: NNC0090-2746 — NNC0090-2746 solution will be self-administered in daily doses of 1.8 mg via SC injection.
  Arms: Treatment Period: NNC0090-2746 QD

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to investigate the efficacy, safety, and tolerability of once-daily subcutaneous (SC) injections of NNC0090-2746 for 12 weeks, as an adjunct to metformin, in participants with T2D.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 70 years, inclusive
* Active diagnosis of T2D for greater than or equal to (>/=) 3 months
* For females of childbearing potential and males with female partners of childbearing potential, agreement to use highly effective contraceptive measures
* Treated with a stable dose of metformin for at least 8 weeks prior to randomization, and expected to remain at the same stable dose throughout study participation
* Hemoglobin A1c (HbA1c) >/= 7.2% and less than or equal to (</=) 10.5%
* Fasting plasma glucose (FPG) less than (<) 250 milligrams per deciliter (mg/dL)
* C-peptide greater than (>) 1.5 nanograms per milliliter (ng/mL)
* Body mass index (BMI) >/= 27 kilograms per meter-squared (kg/m^2) and </= 44 kg/m^2
* Stable weight (+/- 5%) within 12 weeks prior to Screening
* Willing and able to maintain existing diet and exercise habits throughout the study
* Capable of performing SC self-injections on a daily basis during the study

Exclusion Criteria:

* Females who are pregnant or lactating
* History of type 1 diabetes (T1D), diabetes resulting from pancreatic injury, or secondary forms of diabetes such as Cushing's Syndrome or acromegaly
* History of acute metabolic complications such as diabetic ketoacidosis or state of hyperosmolar hyperglycemia
* History of clinically significant diabetic complications such as diabetic proliferative retinopathy or severe diabetic neuropathy (requiring treatment with antidepressants or opioids)
* History of severe hypoglycemia within 6 months prior to Screening
* History of chronic gastrointestinal (GI) conditions that could impede gastric emptying or potentially affect the interpretation of the study data
* History of weight loss surgery or weight loss procedure involving the GI tract, such as gastric bypass, gastric stapling, or gastric banding
* History of an eating disorder (e.g., bulimia, anorexia)
* History of malignancy (except treated basal or squamous cell skin cancer) within 5 years prior to Screening
* Personal or family history of medullary thyroid carcinoma
* History of multiple endocrine neoplasia syndrome type 2
* History of chronic or acute pancreatitis or hemochromatosis
* History of significant cardiovascular disease (such as congestive heart failure New York Heart Association Class II to IV, myocardial infarction within the previous 6 months, coronary disease, or uncontrolled hypertension)
* History of clinically significant renal or liver disease
* History of hypersensitivity or previous intolerance to incretin or glucagon analogues
* Elevations in lipase or amylase levels at Screening > 1.5 times the upper limit of normal (ULN) and considered clinically significant by the investigator
* Positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAG), or hepatitis C antibody test at Screening
* Receipt of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to Screening, or active enrollment in another investigational medication or device study
* Any condition, disorder, or abnormal laboratory test findings at screening that, in the judgment of the investigator, would interfere with the participant's ability to comply with all study requirements, or would require the administration of a treatment during the study that could potentially affect the interpretation of the study data, or would place the participant at unacceptable risk by his/her participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-08-18 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | Day 1; Week 8

SECONDARY OUTCOMES:
Change in body weight | Day 1; Week 8; Week 12
Percent change in body weight | Day 1; Week 8; Week 12
Change in fasting plasma glucose (FPG) | Day 1; Week 12
Change in post-prandial plasma glucose level | Day -7; Week 12
Change in post-prandial insulin level | Day -7; Week 12
Change in post-prandial C-peptide level | Day -7; Week 12
Change in beta-cell function | Day 1; Week 12
  According to the Homeostasis Model Assessment (HOMA) score
Incidence of treatment-emergent adverse events | Day 1; Week 18
Change in percent HbA1c | Day 1; Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (20):
- United States (20):
  - Novo Nordisk Investigational Site, Chino, California
  - Novo Nordisk Investigational Site, Hawaiian Gardens, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Port Orange, Florida
  - Novo Nordisk Investigational Site, Sanford, Florida
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Evanston, Illinois
  - Novo Nordisk Investigational Site, Oxon Hill, Maryland
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Eugene, Oregon
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Manassas, Virginia

REFERENCES:
- [Result] Frias JP, Bastyr EJ 3rd, Vignati L, Tschop MH, Schmitt C, Owen K, Christensen RH, DiMarchi RD. The Sustained Effects of a Dual GIP/GLP-1 Receptor Agonist, NNC0090-2746, in Patients with Type 2 Diabetes. Cell Metab. 2017 Aug 1;26(2):343-352.e2. doi: 10.1016/j.cmet.2017.07.011. PMID 28768173